CLINICAL TRIAL: NCT05962931
Title: Phase I-II, Multicenter, Randomized, Controlled, Proof of Concept Clinical Trial to Determine Feasibility, Safety and Efficacy of the Use of Allogenic Adipose-derived Adult Mesenchymal Stem Cells Expanded on Fibrinhyaluronic Biological Matrix in the Treatment of Venous Ulcer of the Lower Limbs
Brief Title: Clinical Trial With Adipose Tissue Stem Cells on Biological Matrix for the Treatment of Venous Ulcer of the Lower Limbs
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UV/AP/21
Record Dates: First submitted 2023-07-06; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Venous Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bioengineered Artificial Mesenchimal Sheet (BAMS) (Experimental): Allogenic adipose-derived adult mesenchymal stem cells expanded on fibrinhyaluronic biological matrix
  Interventions: Biological: Bioengineered Artificial Mesenchimal Sheet (BAMS)
- Standard treatment (Control) (Active Comparator): Standard treatment
  Interventions: Procedure: Standard treatment (Control)

INTERVENTIONS:
Biological: Bioengineered Artificial Mesenchimal Sheet (BAMS) — Each patient assigned to the experimental treatment group will receive 4 BAMS (1 BAMS/week) at a concentration of about 360,000 cells/cm2.
  Arms: Bioengineered Artificial Mesenchimal Sheet (BAMS)
Procedure: Standard treatment (Control) — Each patient assigned to the control group will undergo a standard treatment procedure for uncomplicated venous ulcers.
  Arms: Standard treatment (Control)

SUMMARY:
Phase I-II, Multicenter, Randomized, Controlled, Proof of Concept Clinical Trial to determine feasibility, safety and efficacy of the use of Allogenic adipose-derived adult mesenchymal stem cells expanded on fibrinhyaluronic biological matrix in the treatment of venous ulcer of the lower limbs.

ELIGIBILITY:
Inclusion Criteria:

1. Signing of the informed consent (IC) after reading the patient information sheet.
2. Over 18 years of both sexes.
3. Active or recurrent venous ulcer in the lower extremity with an area between 5-10 cm2
4. Grade III injury on the Widmer scale.
5. Independence and/or availability to go to the referral center on an outpatient basis.
6. Distal pulses in palpable lower limbs (tibial and foot). ABI between 0.8 - 1.3

Exclusion Criteria:

1. Any pathology for which the investigator considers that compression bandaging is contraindicated and/or previous acute deep vein thrombosis (DVT), within the first 10 days from the onset of symptoms.
2. Grade III obesity with a body mass index (BMI) >40; or underweight patients (BMI <18.5).
3. Active neoplasia and/or being treated with cytostatics.
4. Patients undergoing radiotherapy treatment in areas close to the lesion.
5. Clinical signs of colonization or local infection of the lesion.
6. Patients with more than one lesion compatible with UV in the same lower limb.
7. Erysipelas.
8. Infectious cellulite.
9. Osteomyelitis.
10. Lymphangitis.
11. Chronic lymphedema.
12. Therapy with corticosteroids or immunosuppressants.
13. Venous ulcer grade I or II on the Widmer scale.
14. Lesions close to possible or diagnosed cancerous lesions.
15. Non-localized wounds in the lower extremities.
16. Ongoing infection and/or sepsis.
17. Critical ischemia in the lower limbs or other venous diseases of unknown origin.
18. Immunocompromised patients.
19. Dependent patients with severe mobility limitations.
20. Dialysis patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Factibility of Bioengineered Artificial Mesenchimal Sheet measured as the remission of the treated fistula. | Through study completion, an average of 1 year
  To evaluate the factibility of the topical application of CMTAd in a biological matrix of fibrin-hyaluronic acid on venous ulcers (VU).
Safety of Bioengineered Artificial Mesenchimal Sheet measured by the incidence of adverse events | Through study completion, an average of 1 year
  To examine the safety of cutaneous administration of CMTAd in a biological matrix of fibrin-hyaluronic acid on VUs compared to standard treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Encarnación González Vigil, Principal Investigator — Unidad de A.P. de Atarfe; Mª Ángeles Granado Contrelas, Principal Investigator — Unidad de A.P. de Alfacar; Victor Costela Ruiz, Study Director — Universidad de Granada
Locations (3):
- Spain (3):
  - Unidad de A.P. de Alfacar, Alfacar, Granada
  - Unidad de A.P. de Atarfe, Atarfe, Granada
  - Universidad de Granada, Granada

REFERENCES:
- [Derived] Costela-Ruiz VJ, Gonzalez-Vigil E, Espinosa-Ibanez O, Alcazar-Caballero RM, Melguizo-Rodriguez L, Fernandez-Lopez O, Arias-Santiago S. Application of allogeneic adult mesenchymal stem cells in the treatment of venous ulcers: A phase I/II randomized controlled trial protocol. PLoS One. 2025 May 15;20(5):e0323173. doi: 10.1371/journal.pone.0323173. eCollection 2025. PMID 40373055